CLINICAL TRIAL: NCT01627860
Title: Topiramate in the Treatment of Epilepsy: 1st Add-on vs. Mono-therapy Study in Neuro-Surgical Patients
Brief Title: First Add-on vs. Mono-therapy Study of Topiramate in Neuro-Surgical Patients
Acronym: TEAMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR017248; TOPMATEPY4061 (Other: Janssen-Cilag Taiwan); TOP-TWN-MA4 (Other: Janssen-Cilag Taiwan)
Record Dates: First submitted 2012-05-31; First posted 2012-06-26 (Estimated); Results first posted 2013-05-24 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-09

CONDITIONS: Epilepsy
Keywords: Epilepsy; Topiramate; Neuro-surgical patients; Nervous disorder; Seizures
MeSH Terms: conditions — Epilepsy; Nervous System Diseases; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topiramate add-on therapy (Active Comparator)
  Interventions: Drug: Topiramate add-on therapy
- Topiramate monotherapy (Experimental)
  Interventions: Drug: Topiramate monotherapy

INTERVENTIONS:
Drug: Topiramate add-on therapy — Type=range, unit=mg/day, number=25-200, form=tablet, route=oral use.
  Arms: Topiramate add-on therapy
Drug: Topiramate monotherapy — Type= range, unit= mg/day, number= 25-200, form= tablet, route= oral use.
  Arms: Topiramate monotherapy

SUMMARY:
The purpose of this study is to examine seizure control and tolerability of Topiramate after either transitioning from previous antiepileptic drug (AED) or adding on to previous AED.

DETAILED DESCRIPTION:
This is a multicenter, randomized (treatment is assigned by chance), open-label (everyone who is involved in the trial knows the study drug), parallel group trial. The study has three phases: a retrospective baseline assessment of patients (4 weeks), titration period (8 weeks) and maintenance period (8 weeks). After qualifying for trial entry in the retrospective baseline phase, eligible patients will be randomized in 1:1 ratio to receive either topiramate add-on therapy or topiramate monotherapy. During the titration period (period in which the dose of the study drug is increased or decreased at the discretion of investigator), topiramate, given as morning doses, will be started with daily doses of 25 mg/day for one week. After that, topiramate will be given as morning and evening doses, and the doses will be gradually increased every week to reach the initial target dose of 200 mg/day at the end of titration period. During the maintenance period, the dose of topiramate could be increased or decreased according to the investigator's judgment. Patients should keep seizure diaries during the 16 weeks of topiramate treated period and are followed with once monthly visits to the clinic, at which safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with seizure disorder
* Have been receiving concomitant therapy with one antiepileptic drug (AED), at stable dose prior to trial entry
* Must be dissatisfied with the current treatment

Exclusion Criteria:

* Have treatable cause of seizures (eg, metabolic disturbance, toxic exposure, an active infection, or neoplasm)
* Have grade IV astrocytomas, eg, Glioblastoma multiforme (GBM) or metastases with progression
* Have seizures occurring only in clustered patterns defined as numerous seizures occurring in less than 30 min
* Have had history (within past six months) of a psychiatric or mood disorder requiring electroconvulsive therapy, major tranquilizers, or monoamine oxidase inhibitors
* Have had schizophrenic or history of exhibiting psychotic symptomatology
* Inability to take medication or maintain a seizure calendar, independently or with assistance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Taiwan Clinical Trial, Study Director — Janssen-Cilag Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 55 participants were randomly assigned to receive either topiramate monotherapy or add-on therapy at 6 sites in Taiwan.
Groups:
- Topiramate Monotherapy: Participants received a starting dose of 25 mg/day during week 1 and the dosage increased to 50 mg/day in 2 doses during week 2. Consequently, the dosage increased to 75 mg/day and 100 mg/day in 2 doses during week 3 and week 4, respectively. The dosage increased to 150 mg/day in 2 doses at week 5~6 and 200 mg/day in 2 doses at week 7~8.
- Topiramate add-on Therapy: Participants received topiramate in addition to previous ant-epileptic drug. Participants received a starting dose of 25 mg/day in the morning during week 1 and the dosage was increased to 50 mg/day in 2 doses (morning and evening) during week 2. Consequently, the dosage was increased to 75 mg/day and 100 mg/day in 2 doses during week 3 and week 4, respectively. The dosage was increased to 150 mg/day in 2 doses at week 5~6 and 200 mg/day in 2 doses at week 7~8.
Period: Overall Study
Arm/Group | Topiramate Monotherapy | Topiramate add-on Therapy
Started | 35 | 20
Completed | 23 | 14
Not Completed | 12 | 6
Not completed — Adverse Event | 9 | 4
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Seizure frequency doubled | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate Monotherapy | Topiramate add-on Therapy | Total
Number analyzed (Participants) | 35 | 20 | 55
Age Continuous [Mean (Standard Deviation); unit: years] | 44.1 (11.91) | 42.4 (12.21) | 43.17 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 22 | 13 | 35

OUTCOME MEASURES:

1. Primary Outcome: Seizure Free Rate: Percentage of Participants Who Did Not Have Any Seizure Episode Within the Last Month of the Maintenance Period (ie, Month 4).
Time Frame: Month 4
Population: Intent-To-Treat population: All randomized participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Topiramate Monotherapy | Topiramate add-on Therapy
Number analyzed (Participants) | 35 | 20
Percentage of participants | 88.57 [68.78 to 97.45] | 65.00 [49.20 to 95.34]
Statistical Analysis 1: Comparison: Topiramate Monotherapy vs Topiramate add-on Therapy; Test type: Superiority or Other; p = 0.0759, ANOVA; Difference in Seizure free rate = 23.57, 95% CI 2-sided [-4.21 to 49.00] — Difference in Seizure free rate (Monotherapy minus Add on therapy)

2. Secondary Outcome: Seizure Frequency: Percent Change of Seizure Frequency by the ANCOVA Model During the Month 4
Description: Seizure frequency (seizure count/month) was calculated based on the number of seizure within a month. The mean seizure frequency analyzed by the ANCOVA model at each period.
Time Frame: Baseline (4 weeks retrospective assessment prior to start of titration period) to Month 4
Population: Intent-To-Treat population: All randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Topiramate Monotherapy | Topiramate add-on Therapy
Number analyzed (Participants) | 35 | 20
Percent change | -55.3 (160) | -75.8 (54.1)
Statistical Analysis 1: Comparison: Topiramate Monotherapy vs Topiramate add-on Therapy; Test type: Superiority or Other; p = 0.7102, ANCOVA; Difference in mean percent change = 18.3, 95% CI 2-sided [-81.0 to 117.7] — Difference in mean percent change of seizure frequency (Monotherapy minus Add on therapy)

3. Secondary Outcome: Dosage Administration of Topamax During Month 4
Time Frame: Month 4
Population: Participants who have received study medication during month 4.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Topiramate Monotherapy | Topiramate add-on Therapy
Number analyzed (Participants) | 25 | 14
mg | 182.46 (35.63) | 178.57 (41.98)

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Topiramate Monotherapy | Topiramate add-on Therapy
Serious Adverse Events (participants affected / at risk) | 1/35 | 1/20
Other Adverse Events (participants affected / at risk) | 33/35 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate Monotherapy (N=35) | Topiramate add-on Therapy (N=20)
Herniated Intervertebral Disc (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate Monotherapy (N=35) | Topiramate add-on Therapy (N=20)
Dizziness (Nervous system disorders) | 10 | 4
Headache (Nervous system disorders) | 6 | 3
Hypoaesthesia (Nervous system disorders) | 8 | 1
Decreased appetite (Gastrointestinal disorders) | 5 | 1
Somnolence (Nervous system disorders) | 4 | 2
Weight decreased (Investigations) | 4 | 1
Insomnia (Psychiatric disorders) | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Malaise (General disorders) | 3 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
No limitations were reported in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days